CLINICAL TRIAL: NCT00202202
Title: Survey of the Consultation Service of the Providence Continuing Care Centre Personality Disorder Service Users Satisfaction With the Change in Service Delivery
Brief Title: User Satisfaction Survey - Personality Disorder Service
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PDS001
Record Dates: First submitted 2005-09-09; First posted 2005-09-20 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Borderline Personality Disorder
Keywords: personality disorder; user satisfaction
MeSH Terms: conditions — Borderline Personality Disorder; Personality Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: consultation format

SUMMARY:
Can we improve our community partners satisfaction with a change in how psychiatric consultations are delivered to their clients by our psychiatrist? This survey of users of the service will compare the level of satisfaction before(retrospectively) to after the way the service is provided is changed.

DETAILED DESCRIPTION:
As part of the personality disorder services continuing quality improvement enterprise we sought to review the impact of restructuring on the satisfaction of service community partners with our changed consultation service.

The consultation service was changed as the result of administrative review,part of a larger institution wide process. To review how this change was perceived by agency and individual care providers those who had received consult reports from the last fifty consultations were surveyed about their satisfaction and compared prospectively to the satisfaction of the agencies and individual care providers of clients receiving the next fifty consultations delivered in the new format.

The administrative review had indicated that the consultation reports were unnecessarily comprehensive and in the process time consuming and thereby interfered with timely access to appointments and involved excessive turn around time in the generation of reports. A new streamlined approach using a fill in the blanks type form and brief cover letter and the use of a follow up phone call to the main care giver the same day was devised to address these concerns.

Satisfaction in regards to advice received, length of the report, waiting times for the appointment and for the delivery of the report,legibility and overall satisfaction were surveyed. The satisfaction with telephone feed back was also surveyed.

ELIGIBILITY:
Inclusion Criteria:

* clients referred to the Personality disorder service

Exclusion Criteria:

* self referred clients

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2002-11; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
eight item user satisfaction survey on receipt of the consult report | in the year before and after the change in interview format

SECONDARY OUTCOMES:
demographic factors of the respondents as relate to their satisfaction at time of survey | at the time of suvey completion

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H McNevin, md, Principal Investigator — Queens University
Locations (1):
- Providence Care Mental Health Services, Kingston, Ontario, Canada